CLINICAL TRIAL: NCT00412932
Title: A Prospective, Open Label, Single Arm Study to Evaluation the Safety and Efficacy of an Olmesartan Medoxomil Based Treatment Regimen in Elderly Patients With Hypertension
Brief Title: An Examination of the Blood Pressure Lowering Ability and Safety of Olmesartan Medoxomil in Elderly Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: William Waverczak, Daiichi Sankyo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 866-450
Record Dates: First submitted 2006-12-14; First posted 2006-12-19 (Estimated); Results first posted 2009-09-11 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension
Keywords: Hypertension; Angiotensin Receptor Blocker; Calcium Channel Blocker; Angiotensin Converting Enzyme Inhibitor; Hydrochlorothiazide; Stage I and II Hypertension
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide

INTERVENTIONS:
Drug: Olmesartan medoxomil — Tablets
Drug: Olmesartan medoxomil/hydrochlorothiazide — Tablets

SUMMARY:
This 14 week study will examine the ability of olmesartan medoxomil to lower the blood pressure of patients 65 years of age or older with high blood pressure. The medication being tested has been approved by the FDA for the treatment of high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females greater than 65 years of age
2. Patients with a mean seated systolic blood pressure (MSSBP) greater than or equal to 150 mmHg but less than 200 mm Hg and a mean seated diastolic blood pressure (MSDBP) less than or equal to 109 mmHg following a 2-3 week single blind placebo run-in period.
3. The difference in MSSBP between visits 2 and 3 or between visits 3 and 3x must be less than or equal to 10 mmHg.
4. Patients with a mean daytime (8am-4pm) systolic blood pressure (SBP) greater than or equal to 140 mmHg and less than or equal to 199 mmHg and a mean daytime diastolic blood pressure (DBP) less than or equal to 109 mmHg as measured by an ambulatory blood pressure monitoring device (ABPM) following placebo run-in period.

Exclusion Criteria:

1. History of stroke or transient ischemic attack (TIA) within the last one year.
2. History of myocardial infarction, angina, coronary angioplasty, coronary artery bypass graft, or heart failure within the past 6 months.
3. Severe hypertension (diastolic blood pressure greater than 115 mmHg or systolic blood pressure greater than or equal to 200 mmHg).
4. Patients with secondary hypertension of any etiology, such as renal disease, pheochromocytoma or Cushing's syndrome.
5. Type I diabetes or Type II diabetics not on stable treatment for greater than or equal to 4 weeks and plasma glucose greater than 160 mg/dl.
6. Evidence of symptomatic resting bradycardia, congestive heart failure, or hemodynamically significant cardiac valvular disease.
7. Presence of heart block greater than first degree sinoatrial block, Wolff-Parkinson-White Syndrome, Sick Sinus Syndrome, an accessory bypass tract, atrial fibrillation, atrial flutter or any arrhythmia requiring medication.
8. Serum Creatinine greater than 1.7 mg/dl, or other abnormal laboratory values deemed clinically significant by the investigator.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 178 (Actual)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Long Beach, California
  - Los Angeles, California
  - Pomona, California
  - Roseville, California
  - Tustin, California
  - Farmington, Connecticut
  - Jupiter, Florida
  - Lauderdale Lakes, Florida
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - Chicago, Illinois
  - Wichita, Kansas
  - Madisonville, Kentucky
  - Auburn, Maine
  - Baltimore, Maryland
  - Oxon Hill, Maryland
  - Florissant, Missouri
  - Berlin, New Jersey
  - Williamsville, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Greer, South Carolina
  - Corpus Christi, Texas
  - Richardson, Texas
  - Norfolk, Virginia
  - Madison, Wisconsin

REFERENCES:
- [Derived] Germino FW, Neutel JM, Dubiel R, Maa JF, Chavanu KJ. Efficacy of olmesartan medoxomil and hydrochlorothiazide fixed-dose combination therapy in patients aged 65 years and older with stage 1 and 2 hypertension or isolated systolic hypertension. Am J Cardiovasc Drugs. 2012 Oct 1;12(5):325-33. doi: 10.1007/BF03261841. PMID 22920048
- [Derived] Neutel J, Kereiakes DJ, Stoakes KA, Maa JF, Shojaee A, Waverczak WF. Blood pressure-lowering efficacy of an olmesartan medoxomil/hydrochlorothiazide-based treatment algorithm in elderly patients (age >/=65 years) stratified by age, sex and race: subgroup analysis of a 12-week, open-label, single-arm, dose-titration study. Drugs Aging. 2011 Jun 1;28(6):477-90. doi: 10.2165/11589460-000000000-00000. PMID 21639407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 37 US sites (private medical practices and small clinics) over 13 months (Nov 29,06 to Dec 28,07) from each physician's clientele base. Approximately 200 eligible participants, men and women at least 65 years of age with hypertension or uncontrolled hypertension on current medication, were to receive active treatment
Pre-assignment Details: After 3-4 weeks of placebo, patients with a systolic pressure (SBP) ≥150 ≤199mmHg and diastolic pressure (DBP) ≤109 mmHg at the last 2 visits, and 8-hr daytime SBP >140 and ≤199 mmHg and DBP ≤109 mmHg by ambulatory blood pressure monitoring were entered.All started with Olmesartan 20 mg and were titrated if their blood pressure was not controlled
Groups:
- Active Treatment Period: All participants started this arm with 20 mg olmesartan medoxomil (Olm). After 3 weeks participants were titrated to 40g Olm, if their blood pressure was not controlled. After 6 weeks they were titrated to the next step which now included Olm 40 mg + hydrochlorothiazide (HCTZ) 12.5 mg if their blood pressure was not controlled. After 9 weeks they were titrated to the next step which now included Olm 40 mg + HCTZ 25 mg if their blood pressure was not controlled.
Period: Olmesartan (Olm) 20 mg
Arm/Group | Active Treatment Period
Started | 178
Completed | 171
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Other | 1
Period: Olmesartan 40 mg
Arm/Group | Active Treatment Period
Started | 169 (171 -1 met blood pressure goal (stayed on olmesartan 20) -1 who erroneously skipped this step = 169.)
Completed | 161
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 1
Period: Olm+Hydrochlorothiazide 12.5 mg
Arm/Group | Active Treatment Period
Started | 159 (161 -2 met blood pressure goal (stayed on olmesartan 40) = 159)
Completed | 153
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3
Period: Olm+ Hydrochlorothiazide 25 mg
Arm/Group | Active Treatment Period
Started | 125 (153 -28 met their blood pressure goal (stayed on olmesartan 40/hydrochlorothiazide 12.5) = 125)
Completed | 123
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment Period: All participants started the active treatment period with 20 mg olmesartan medoxomil (Olm). After 3 weeks participants were titrated to 40 mg Olm, if their blood pressure was not controlled. After 6 weeks they were titrated to the next step which now included Olm 40 mg + hydrochlorothiazide (HCTZ) 12.5 mg if their blood pressure was not controlled. After 9 weeks they were titrated to the next step which now included Olm 40 mg + HCTZ 25 mg if their blood pressure was not controlled.
Arm/Group | Active Treatment Period
Number analyzed (Participants) | 178
Age Continuous [Mean (Standard Deviation); unit: years] | 72.0 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 93
Region of Enrollment [Number; unit: participants]
  United States | 178
Baseline stage of hypertension [Number; unit: participants] — Stage I hypertension is defined as systolic blood pressure (SBP) of 140 - 159 mmHg and diastolic blood pressure (DBP) of 90 - 99 mmHg; Stage II is defined as SBP ≥ 160 mmHg or DBP ≥ 100 mm Hg.
  participants
    Stage 1 hypertension | 62
    Stage 2 hypertension | 116
Baseline 24-hour ambulatory diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 80.7 (8.5)
Baseline 24-hour ambulatory systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 149.1 (11.2)
Baseline diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 87.7 (9.6)
Baseline heart rate [Mean (Standard Deviation); unit: beats/minute] | 71.5 (11.4)
Baseline systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 165.5 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean 24-hour Ambulatory Systolic Blood Pressure After 12 Weeks of Active Treatment
Description: All participants started the treatment arm with 20 mg olmesartan medoxomil (Olm). If their blood pressure was not controlled, participants were titrated at 3-week intervals to: Olm 40 mg, then, if needed Olm 40 mg + hydrochlorothiazide (HCTZ) 12.5 mg, then, if needed Olm 40 mg + HCTZ 25 mg This outcome measure included all participants at the end of the 12-week treatment period regardless of whether or not they were titrated. They had to have both baseline and 12-week ambulatory blood pressure measurements.
Time Frame: baseline to 12 weeks
Population: 178 participants started the active treatment period. 23 dropped out. 150=The ambulatory blood pressure monitoring (ABPM) subset was defined as subjects who received at least one dose of active study medication and had a baseline and week 12 ABPM.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study
Number analyzed (Participants) | 150
mm Hg | -25.7 (0.96)
Statistical Analysis 1: Comparison: Overall Study; The sample size of this study was not based on the statistical power consideration and was considered as sufficient for the evaluation of the efficacy and safety of the proposed olmesartan medoxomil-based treatment regimen; Test type: Superiority or Other; p < 0.0001, one-sample t-test — No multiplicity adjustments

2. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Diastolic Blood Pressure After 12 Weeks of Active Treatment.
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study
Number analyzed (Participants) | 150
mm Hg | -12.3 (0.55)
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p < 0.0001, One-sample t-test

3. Secondary Outcome: Change From Baseline in Mean Daytime (8am-4pm) and Mean Nighttime (10pm-6am)Ambulatory Systolic Blood Pressure After 12 Weeks of Active Treatment
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study
Number analyzed (Participants) | 150
mm Hg
  Daytime | -26.5 (1.10)
  Nighttime | -24.4 (1.04)
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p < 0.0001, one-sample t-test — No multiplicity adjustments. This P-Value applies to both the daytime and nighttime periods

4. Secondary Outcome: Change From Baseline in Mean Daytime (8am-4pm) and Mean Nighttime (10 Pm-6am) Ambulatory Blood Pressure Monitored Diastolic Blood Pressure After 12 Weeks of Active Treatment
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Population: 178 participants started the active treatment period. 23 dropped out. 150=The ambulatory blood pressure monitoring (ABPM) subset was defined as subjects who received at least one dose of active study medication and had baseline and week 12 ABPM measurements.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study
Number analyzed (Participants) | 150
mm Hg
  Daytime | -13.0 (0.65)
  Nighttime | -11.5 (0.60)
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p < 0.0001, one-sample t-test — No multiplicity adjustments. The P-Value of <0.0001 applies to both daytime and nighttime periods

5. Secondary Outcome: Number of Subjects Who Achieved Mean 24-hour Ambluatory Blood Pressure of <140/90 mm Hg, Systolic Blood Pressure <140 mm Hg, and Diastolic Blood Pressure <90 mm Hg After 12 Weeks of Active Treatment
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Overall Study
Number analyzed (Participants) | 150
participants
  BP<140/90 mm Hg | 133
  SBP<140 mm Hg | 133
  DBP<90 mm Hg | 149

6. Secondary Outcome: Number of Subjects Who Achieved Mean Daytime (8am - 4pm) Ambulatory Blood Pressure of <140/90 mm Hg, Systolic Blood Pressure <140 mm Hg, and Diastolic Blood Pressure <90 mm Hg After 12 Weeks of Active Treatment.
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Overall Study
Number analyzed (Participants) | 150
participants
  BP<140/90 mm Hg | 120
  SBP<140 mm Hg | 120
  DBP<90 mm Hg | 145

7. Secondary Outcome: Number of Subjects Who Achieved Mean Nighttime (10pm - 6am) Ambulatory Blood Pressure of <140/90 mm Hg, Systolic Blood Pressure <140 mm Hg, and Diastolic Blood Pressure <90 mm Hg After 12 Weeks of Active Treatment.
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Overall Study
Number analyzed (Participants) | 150
participants
  BP<140/90 mm Hg | 143
  SBP<140 mm Hg | 143
  DBP<90 mm Hg | 149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"If identified by Daiichi Sankyo, Inc. (DSI), any of DSI's confidential information as defined herein shall be deleted. Nothing in this Publication section shall be taken as giving DSI the right of editorial control over any publication prepared by the study site."